CLINICAL TRIAL: NCT06400706
Title: Effect of Electroencephalography (SEF and PSI) Guided General Anesthesia on Postoperative Delirium and Anesthetic Consumption in Children Underwent Dental Rehabilitation: A Randomized Controlled Trial
Brief Title: Effect of Electroencephalography Guided General Anesthesia on Postoperative Delirium in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ozlem Kocaturk, Prof. Dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AADUDHF 2023/34
Record Dates: First submitted 2024-04-21; First posted 2024-05-06 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Delirium; Postoperative Pain
Keywords: General anesthesia; Electroensephalography; Emergence delirium
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEG Group (Experimental): EEG guided general anesthesia: General anesthesia is guided by SedLine (EEG-guided care). The goal of EEG-guided care is to maintain spectral edge frequency (SEF) between 10 and 15 and patient state index (PSI) between 25 and 50.
  Interventions: Procedure: EEG guided general anesthesia
- Control (No Intervention): Standard general anesthesia: Anesthesia management is performed to keep the minimal alveolar concentration (MAC) value at 0.9 and intraoperative drug use is adjusted according to the experience of the anesthesiologist.

INTERVENTIONS:
Procedure: EEG guided general anesthesia — EEG guided general anesthesia: General anesthesia is guided by SedLine (EEG-guided care). The goal of EEG-guided care is to maintain spectral edge frequency (SEF) between 10 and 15 and patient state index (PSI) between 25 and 50.
  Arms: EEG Group

SUMMARY:
Participants aged 4-10 years (92 patients), who came to the Hospital Operating Room at the University Faculty of Dentistry with an indication for dental treatment under general anesthesia due to lack of cooperation, will be selected by simple randomization and divided into 2 groups. One group of participants who will undergo routine general anesthesia and dental treatment procedures will receive routine monitoring (Group I), and the other group will receive EEG monitoring (Group II) in addition to routine monitoring. Electrocardiography (ECG), oxygen saturation (SpO2), non-invasive blood pressure (NIBP), endtidal carbon dioxide (EtCO2), endtidal sevoflurane (EtSev) parameters observed as routine monitoring of the patients will be recorded and the minimal alveolar concentration (MAC) value will be kept at 0.9. Anesthesia management will be performed, and in Group II, in addition to routine monitoring, anesthesia management will be carried out to keep the SEF values observed in the EEG between 10-15 and PSI values between 25-50. Routine general anesthesia procedures and dental treatments will not differ between groups.

Age, gender, weight, intubation type, ASA, previous surgical experience, anesthesia duration, number of extracted teeth with decayed fillings (dmft) values will also be recorded.

In the intraoperative period; hemodynamic parameters (average heart rate, blood pressure and oxygen saturation values) and amounts of medication consumed (most tidal sevoflurane percentages in induction and maintenance, presence of burst suppression, sevoflurane/fentanyl/rocuronium consumption). The participants, whose operation is completed, will be taken to the recovery room and any post-operative discomfort will be noted. The cases will be recorded in the report form.

In the postoperative period; Extubation time, agitation (PAED scores) and pain (FLACC, VAS-ORF) scores will be recorded during extubation and 10, 20, 30 minutes and 2 hours after extubation, and recovery time, hospital stay, presence of nausea and vomiting will also be recorded.

Modified Aldrete Recovery Score (MAS) will be used for recovery criteria and MAS >8 will be considered as a recovery indicator. The Pediatric Anesthesia Early Delirium Scale (PAED) will be used to evaluate early agitation. FLACC and VAS-ORF scale will be used as pain scales.

DETAILED DESCRIPTION:
Postoperative delirium (POD) is an acute postoperative behavioral change defined as an impairment in the child's awareness or attention to the environment, accompanied by disorientation and perceptual changes, including hypersensitivity to stimuli and hyperactive motor behavior, usually in the immediate post-anesthesia period. The incidence of POD may depend largely on age, anesthesia technique, surgical procedure, and adjunctive medication administration. Its incidence in preschool children receiving sevoflurane anesthesia varies between 10-80%. Although POD is mostly self-limiting and occurs within the first minutes of the postoperative period, physical injuries cannot be ignored as children can move their limbs uncontrollably, get rid of their catheters, and even lose important equipment.

Prevention of POD includes pharmacological treatment and non-pharmacological treatment. Pharmacological treatment, including the administration of midazolam, ketamine, dexmedetomidine, and melatonin in the preoperative or intraoperative period, is effective, but these measures can prolong the stay in the postoperative anesthesia care unit (PACU) and cause many adverse reactions, such as postoperative nausea and vomiting, respiratory depression. Non-pharmacological treatments, such as parental companionship, preoperative education, or playing music upon entering the room, offer therapeutic effects at lower cost and greater convenience. Therefore, finding ways to prevent POD using non-pharmacological treatments is valuable.

Nowadays, more and more anesthesiologists titrate the anesthesia dose by monitoring the depth of anesthesia. In 2020, electroencephalography (EEG) monitoring was recommended by the American Society of Anesthesiologists (ASA) as one of the important organ monitoring methods to guide general anesthesia management. In the adult population, the potential benefits of monitoring intraoperative depth of anesthesia have been confirmed, including a lower incidence of hypotension under anesthesia and intraoperative awareness, faster awakening and recovery time, and reduced drug dosage use. Many meta-analyses have shown that anesthesia management through EEG monitoring can reduce the occurrence of POD in adult patients undergoing general anesthesia. EEG and depth of anesthesia monitoring have been used in pediatric anesthesia management since 2000; It is especially recommended for use in children who have undergone major or long-term surgery. EEG monitoring in pediatric anesthesia has been proven to be beneficial for children by reducing anesthetic consumption. Pediatric routine anesthesia management largely depends on the experience of the anesthesiologist.

Xu et al. reported that in pediatric surgery, EEG parameters [SEF (spectral edge frequency), PSI (patient state index), DSA (density spectral array) and raw EEG waves] may be more effective than special indices in reflecting the depth of anesthesia. Recent studies have also reported that SEF may be more effective in representing the depth of anesthesia, and that DSA can be used as a measure of the depth of anesthesia in young children undergoing sevoflurane anesthesia. In addition, in the studies of Koch et al., raw EEG features were analyzed in children undergoing general anesthesia and some relationships were found between POD and EEG epileptiform discharges. However, it is still unclear whether the use of these EEG parameters (SEF, DSA, raw EEG wave) can reduce the incidence of POD.

In this study, the investigators used SEF, PSI, DSA and EEG waves to monitor the depth of anesthesia in children. SEF, PSI, DSA and raw EEG waves can reflect the depth of anesthesia more precisely. The aim is to investigate whether the use of SEF, DSA and EEG wave measurement to guide and manage pediatric anesthesia can reduce the incidence of POD and anesthesia consumption.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II,
* Those who will undergo elective dental procedures under general anesthesia
* Cases where anesthesia duration will be more than 1 hour

Exclusion Criteria:

* Having a history of serious neurological or mental illness
* Having growth-developmental retardation
* Parents or children do not want to participate in the study or are participating in another research study at the same time.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Emergence Delirium | From date of randomization until the date of first documented progression (up to thirty weeks)
  It is measured with the Pediatric Anesthesia Emergency Delirium Scale (PAEDS). The higher the score, the more severe the child's agitation; Scores > 2 indicate postoperative agitation, scores > 10 indicate postoperative delirium.

SECONDARY OUTCOMES:
Anesthetic Consumption | From date of randomization until the date of first documented progression (up to thirty weeks)
  Sevoflurane/Fentanyl/Rocuronium consumption during surgery
Postoperative Pain | From date of randomization until the date of first documented progression (up to thirty weeks)
  FLACC scale will be used as pain scales. The highest score is 10. The more severe the child's pain, the higher the score.
Postoperative Discomfort | From date of randomization until the date of first documented progression (up to thirty weeks
  VAS-ORF scale will be used as pain scales. The highest score is 10. The more severe the child's pain, the higher the score.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Kocaturk, MD, Prof., Study Director — Adnan Menderes University Faculty Of Dentistry Division Of Anesthesiology
Locations (1):
- Aydın Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang CJ, Jin Z, Sands LP, Pleasants D, Tabatabai S, Hong Y, Leung JM. ADAPT-2: A Randomized Clinical Trial to Reduce Intraoperative EEG Suppression in Older Surgical Patients Undergoing Major Noncardiac Surgery. Anesth Analg. 2020 Oct;131(4):1228-1236. doi: 10.1213/ANE.0000000000004713. PMID 32925344
- [Result] Han Y, Miao M, Li P, Yang Y, Zhang H, Zhang B, Sun M, Zhang J. EEG-Parameter-Guided Anesthesia for Prevention of Emergence Delirium in Children. Brain Sci. 2022 Sep 5;12(9):1195. doi: 10.3390/brainsci12091195. PMID 36138931
- [Result] Sumner M, Deng C, Evered L, Frampton C, Leslie K, Short T, Campbell D. Processed electroencephalography-guided general anaesthesia to reduce postoperative delirium: a systematic review and meta-analysis. Br J Anaesth. 2023 Feb;130(2):e243-e253. doi: 10.1016/j.bja.2022.01.006. Epub 2022 Feb 17. PMID 35183345